CLINICAL TRIAL: NCT06461052
Title: Information and Music Therapy as a Means of Reducing Preoperative Anxiety in Outpatient Surgery. Outpatient Surgery: a Before-and-after Study
Brief Title: Information and Music Therapy as a Means of Reducing Preoperative Anxiety in Outpatient Surgery.
Acronym: Harmonie
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021_0188; 2023-A02493-42 (Registry Identifier: ID-RCB number)
Record Dates: First submitted 2024-05-24; First posted 2024-06-14 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Ambulatory Surgery
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Prospective study, parallel group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): patient information via a video explaining the procedure, followed by a15-minute music therapy session of your choice in the OR waiting room.
  Interventions: Procedure: music therapy

INTERVENTIONS:
Procedure: music therapy — The patient will benefit from viewing the video and the music therapy session in the waiting room of the operating room. The patient will be asked again for their anxiety score using an anxiety scale. This will define the main outcome of the study. Following this collection and in order not to influence the response, investigators will collect from the patient his compliance with the two proposed techniques as well as his appreciation of the tool.
  Arms: Intervention

SUMMARY:
This is a monocentric, prospective, before-and-after, open-label controlled study, two groups of 99 patients each: "control" group - usual care - versus "intervention" group "Intervention" group - patient information via an explanatory video followed by a 15-minute music therapy session of the patient's choice in the operating waiting room.

DETAILED DESCRIPTION:
Although general anaesthesia is used for almost 10 million procedures a year, and the safety of this procedure has improved considerably over the last 25 years, notably with the "safety decree" of December 1994, general anaesthesia remains deeply associated with high levels of preoperative anxiety. Anxiety levels are correlated with two perioperative factors:

* the need for more anesthetic agents to achieve the same level of depth of anesthesia in anxious patients compared to non-anxious/low-anxiety patients
* Development of chronic postoperative pain.

The preoperative consultation and visit by an anaesthetist is an important meeting point to reduce these high levels of anxiety. On the other hand, systematic benzodiazepine-based premedication has been abandoned for some years now, and taking action to reduce the level of anxiety is one of today's challenges, using a variety of means: organizational, video, music, virtual reality, hypnosis...

Unfortunately, the level of publication on the subject remains low.

Currently, a local analysis of this pathway shows several waiting times for which patients are not necessarily informed, and which can generate anxiety during treatment. In addition, our preliminary survey on the subject showed a specific need for information on pain management and anaesthesia recovery. and anesthesia recovery.

The goal of this study was to design a two-group comparative study aiming of significantly reducing perioperative anxiety in outpatients by implementing simple solutions. More specifically, our project focuses on the impact of music therapy and dedicated information via an explanatory video of the patient's journey through the operating room on the level of perioperative anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Any patient over the age of 18 undergoing scheduled outpatient surgery in the central
* under general anesthesia. The surgeries surgeries concerned are versatile: Digestive (inguinal hernias, proctology, cholecystectomy, etc.), thoracic endoscopy (biopsy examination under GA), gynecological (hysteroscopy, diagnostic laparoscopy diagnostic laparoscopy, cerclage...), ENT (endoscopies, septoplasty, meatotomy...), Urology (JJ catheter insertionTOT/TVT, botulinum toxin injection...), vascular (stripping)
* Patient with oral non-opposition prior to any study procedure
* Not to have objected to inclusion in the research
* Patient affiliated to a health insurance scheme

Exclusion Criteria:

* Patients undergoing emergency surgery, considered full stomach
* Patient not respecting the central block route (interventional radiology in this case)
* First patients in the program because they present the risk of less than than 15 minutes
* Patients who do not understand French
* Patient deprived of liberty or under guardianship
* Pregnant or breast-feeding women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-07-05 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Compare the proportion of patients with high anxiety (Visual Analog Score (VAS) for pain greater than or equal to 40/100) in operating waiting room between the two groups (before and after implementation of the actions). | up to 24 hours
  The primary endpoint was the presence or absence of high anxiety in operating waiting room (T2), measured by an VAS score > 40/100. A range of scores from 0-100. A higher score indicates greater pain intensity.

SECONDARY OUTCOMES:
Compare anxiety levels in preoperative reception unit (T1) and in post anesthesia care unit room (T3) between the two groups: Amsterdam Preoperative Anxiety and Information Scale (APAIS) and VAS score | up to 24 hours
  VAS score and APAIS in preoperative reception unit (T1) and in post anesthesia care unit room (T3). A range of scores from 0-100. A higher score indicates greater pain intensity. The APAIS scale is a six-item questionnaire graded on a five-point Likert scale from 1=not at all to 5=extremely
Compare anxiety levels in operating waiting room (T2) | up to 24 hours
  VAS score in operating room waiting room (T2). A range of scores from 0-100. A higher score indicates greater pain intensity.
Compare the time to loss of consciousness measured in the operating room between both groups | up to 24 hours
  Time to loss of consciousness measured in the operating room (time between injection of hypnotic agent (propofol) and a sleep depth measurement less than 60)
Compare the amount of propofol (mg/kg) at induction required to achieve loss of consciousness between the two groups. | up to 24 hours
  Amount of propofol (mg/kg) at induction required to achieve loss of consciousness
Evaluate the level of satisfaction of each action implemented using a specific questionnaire at the end of the program. | up to 24 hours
  Level of satisfaction using a specific questionnaire at the end of the Licker scale
Evaluate the proportion of dropouts for each action, i.e. the proportion of patients who did not viewed the video until the end, or did not complete the entire music therapy session. | up to 24 hours
  Action completed in full or partially yes or no

CONTACTS AND LOCATIONS:
Overall Officials: Morgan LE GUEN, MD, Principal Investigator — FOCH Hospital
Locations (2):
- France (2):
  - DRCI FOCH Hospital, Suresnes
  - FOCH Hospital, Suresnes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedrich S, Reis S, Meybohm P, Kranke P. Preoperative anxiety. Curr Opin Anaesthesiol. 2022 Dec 1;35(6):674-678. doi: 10.1097/ACO.0000000000001186. Epub 2022 Sep 21. PMID 36131642
- [Background] Maurice-Szamburski A, Auquier P, Viarre-Oreal V, Cuvillon P, Carles M, Ripart J, Honore S, Triglia T, Loundou A, Leone M, Bruder N; PremedX Study Investigators. Effect of sedative premedication on patient experience after general anesthesia: a randomized clinical trial. JAMA. 2015 Mar 3;313(9):916-25. doi: 10.1001/jama.2015.1108. PMID 25734733
- [Background] Eijlers R, Dierckx B, Staals LM, Berghmans JM, van der Schroeff MP, Strabbing EM, Wijnen RMH, Hillegers MHJ, Legerstee JS, Utens EMWJ. Virtual reality exposure before elective day care surgery to reduce anxiety and pain in children: A randomised controlled trial. Eur J Anaesthesiol. 2019 Oct;36(10):728-737. doi: 10.1097/EJA.0000000000001059. PMID 31356373
- [Background] Gurler H, Yilmaz M, Turk KE. Preoperative Anxiety Levels in Surgical Patients: A Comparison of Three Different Scale Scores. J Perianesth Nurs. 2022 Feb;37(1):69-74. doi: 10.1016/j.jopan.2021.05.013. Epub 2021 Nov 19. PMID 34810072
- [Background] Hedayati J, Bagheri-Nesami M, Elyasi F, Hosseinnataj A. The Effect of Music Therapy on the Pain and Anxiety Levels of Patients Experiencing Wound Healing by Suturing in the Emergency Wards. Anesth Pain Med. 2023 Feb 25;13(1):e132943. doi: 10.5812/aapm-132943. eCollection 2023 Feb. PMID 37409003
- [Background] Maurice-Szamburski A, Loundou A, Capdevila X, Bruder N, Auquier P. Validation of the French version of the Amsterdam preoperative anxiety and information scale (APAIS). Health Qual Life Outcomes. 2013 Oct 7;11:166. doi: 10.1186/1477-7525-11-166. PMID 24099176
- [Background] Celik F, Edipoglu IS. Evaluation of preoperative anxiety and fear of anesthesia using APAIS score. Eur J Med Res. 2018 Sep 11;23(1):41. doi: 10.1186/s40001-018-0339-4. PMID 30205837
- [Background] Eberhart L, Aust H, Schuster M, Sturm T, Gehling M, Euteneuer F, Rusch D. Preoperative anxiety in adults - a cross-sectional study on specific fears and risk factors. BMC Psychiatry. 2020 Mar 30;20(1):140. doi: 10.1186/s12888-020-02552-w. PMID 32228525